CLINICAL TRIAL: NCT05979454
Title: Value of Krebs Von Den Lungen-6 Assay in Rheumatoid Artheritis-associated Interstitial Lung Disease
Brief Title: Value of KL-6 in Rheumatoid Arthritis-Associated ILD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Safaa Abd El-gayed Eid, Principal investigator, Assiut University
Other Study IDs: ABBAAS
Record Dates: First submitted 2023-07-28; First posted 2023-08-07 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-11

CONDITIONS: Rheumatoid Arthritis-Associated Interstitial Lung Disease
MeSH Terms: interventions — Spirometry

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum sample
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rheumatoid Arthritis-associated Interstitial Lung Disease: Krebs von den Lungen-6 (KL6)
  Interventions: Diagnostic Test: Krebs von den Lungen-6 (KL6)

INTERVENTIONS:
Diagnostic Test: Krebs von den Lungen-6 (KL6) — KL-6 concentration will be measured using Sandwich ELISA technique (SinoGene Clone Biotech, China).
  Other Names: Spirometry; HRCT Chest

SUMMARY:
Evaluation of serum KL6 level in rheumatoid arthritis-associated interstitial lung disease (RA-ILD).

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is one of the most common connective tissue diseases (CTD). Its prevalence is increasing worldwide . It is responsible for a considerable number of hospital visits in Egyptian Hospitals . Pumlonary involvement is common in rheumatoid arthritis (RA). Interstitial lung disease associated rheumatoid arthritis (ILD-RA) is responsible for significant morbidity and mortality .

Krebs von den Lungen 6 (KL-6) is a mucin like glycoprotein that is found mainly on the surface of type II pneumocytes as well as in bronchiolar epithelial cells . It has chemotactic and anti-apoptotic action on fibroblasts , hence, it is considered as a marker of pulmonary epithelial cell injury .

Krebs von den Lungen-6 (KL6) has been found to be a valuable diagnostic tool in many interstitial lung diseases. KL6 was found to be a valuable prognostic marker, as well as a marker for disease severity in idiopathic pulmonary fibrosis (IPF) . KL6 was found useful as well in predicting in-hospital mortality in patients with Acute exacerbation of interstitial lung disease (AE-ILD) . KL-6 serum level can serve as a diagnostic marker for connective tissue disease-associated interstitial lung disease (CTD-ILD). It can be used to monitor effectiveness of medical treatment and patient response to pulse therapy . Its value in Rheumatoid Arthritis-associated Interstitial Lung Disease (RA-ILD) has not yet been adequately investigated.

ELIGIBILITY:
Diagnosis of RA will be based on American College of Rheumatology/European League against Rheumatism (ACR-EULAR) classification criteria 2010.

Inclusion Criteria:

* all patients have rheumatoid arthritis-associated interstitial lung disease

Exclusion Criteria:

* Patients with any evidence of infection will be excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients have rheumatoid arthritis-associated interstitial lung disease
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
KL-6 | one day
  detect its serum level

SECONDARY OUTCOMES:
Spirometry | one day
  FEV1, FVC, FVC/FEV1 will be measured.
HRCT chest | one day
  It will be will be assessed by the radiologist to determine pulmonary involvement.

CONTACTS AND LOCATIONS:
Overall Officials: Safaa A Eid, Fellow, Principal Investigator — Assiut University
Locations (1):
- Safaa A Eid, Asyut, Egypt

REFERENCES:
- [Background] Finckh A, Gilbert B, Hodkinson B, Bae SC, Thomas R, Deane KD, Alpizar-Rodriguez D, Lauper K. Global epidemiology of rheumatoid arthritis. Nat Rev Rheumatol. 2022 Oct;18(10):591-602. doi: 10.1038/s41584-022-00827-y. Epub 2022 Sep 6. PMID 36068354
- [Background] Sakr BR, Elfishawi MM, ElArousy MH, Hatw AK, AbdulKarim AN, Tammam AB, Kotp AN, Hamed ME, Genedy IE, Desouky EDE, Nawito ZO. Rheumatoid arthritis: A single-center Egyptian experience. Immunol Invest. 2018 Apr;47(3):293-302. doi: 10.1080/08820139.2018.1425700. Epub 2018 Jan 16. PMID 29336618
- [Background] Olson AL, Swigris JJ, Sprunger DB, Fischer A, Fernandez-Perez ER, Solomon J, Murphy J, Cohen M, Raghu G, Brown KK. Rheumatoid arthritis-interstitial lung disease-associated mortality. Am J Respir Crit Care Med. 2011 Feb 1;183(3):372-8. doi: 10.1164/rccm.201004-0622OC. Epub 2010 Sep 17. PMID 20851924
- [Background] Doyle TJ, Lee JS, Dellaripa PF, Lederer JA, Matteson EL, Fischer A, Ascherman DP, Glassberg MK, Ryu JH, Danoff SK, Brown KK, Collard HR, Rosas IO. A roadmap to promote clinical and translational research in rheumatoid arthritis-associated interstitial lung disease. Chest. 2014 Mar 1;145(3):454-463. doi: 10.1378/chest.13-2408. PMID 24590021
- [Background] Kohno N, Inoue Y, Hamada H, Fujioka S, Fujino S, Yokoyama A, Hiwada K, Ueda N, Akiyama M. Difference in sero-diagnostic values among KL-6-associated mucins classified as cluster 9. Int J Cancer Suppl. 1994;8:81-3. doi: 10.1002/ijc.2910570717. PMID 8194900
- [Background] Hirasawa Y, Kohno N, Yokoyama A, Inoue Y, Abe M, Hiwada K. KL-6, a human MUC1 mucin, is chemotactic for human fibroblasts. Am J Respir Cell Mol Biol. 1997 Oct;17(4):501-7. doi: 10.1165/ajrcmb.17.4.2253. PMID 9376125
- [Background] Arnold DT, Donald C, Lyon M, Hamilton FW, Morley AJ, Attwood M, Dipper A, Barratt SL. Krebs von den Lungen 6 (KL-6) as a marker for disease severity and persistent radiological abnormalities following COVID-19 infection at 12 weeks. PLoS One. 2021 Apr 29;16(4):e0249607. doi: 10.1371/journal.pone.0249607. eCollection 2021. PMID 33914762
- [Background] Jiang D, Xiao H, Dong R, Geng J, Xie B, Ren Y, Dai H. Krebs von den Lungen-6 levels in untreated idiopathic pulmonary fibrosis. Clin Respir J. 2022 Mar;16(3):234-243. doi: 10.1111/crj.13475. Epub 2022 Jan 26. PMID 35081277
- [Background] Choi MG, Choi SM, Lee JH, Yoon JK, Song JW. Changes in blood Krebs von den Lungen-6 predict the mortality of patients with acute exacerbation of interstitial lung disease. Sci Rep. 2022 Mar 22;12(1):4916. doi: 10.1038/s41598-022-08965-9. PMID 35318424
- [Background] Ma H, Lu J, Song Y, Wang H, Yin S. The value of serum Krebs von den lungen-6 as a diagnostic marker in connective tissue disease associated with interstitial lung disease. BMC Pulm Med. 2020 Jan 8;20(1):6. doi: 10.1186/s12890-019-1043-z. PMID 31915006
- [Background] Aletaha D, Neogi T, Silman AJ, Funovits J, Felson DT, Bingham CO 3rd, Birnbaum NS, Burmester GR, Bykerk VP, Cohen MD, Combe B, Costenbader KH, Dougados M, Emery P, Ferraccioli G, Hazes JM, Hobbs K, Huizinga TW, Kavanaugh A, Kay J, Kvien TK, Laing T, Mease P, Menard HA, Moreland LW, Naden RL, Pincus T, Smolen JS, Stanislawska-Biernat E, Symmons D, Tak PP, Upchurch KS, Vencovsky J, Wolfe F, Hawker G. 2010 Rheumatoid arthritis classification criteria: an American College of Rheumatology/European League Against Rheumatism collaborative initiative. Arthritis Rheum. 2010 Sep;62(9):2569-81. doi: 10.1002/art.27584. PMID 20872595
- [Background] Graham BL, Steenbruggen I, Miller MR, Barjaktarevic IZ, Cooper BG, Hall GL, Hallstrand TS, Kaminsky DA, McCarthy K, McCormack MC, Oropez CE, Rosenfeld M, Stanojevic S, Swanney MP, Thompson BR. Standardization of Spirometry 2019 Update. An Official American Thoracic Society and European Respiratory Society Technical Statement. Am J Respir Crit Care Med. 2019 Oct 15;200(8):e70-e88. doi: 10.1164/rccm.201908-1590ST. PMID 31613151